CLINICAL TRIAL: NCT00422630
Title: Dietary Interventions for Insulin Resistance and the Metabolic Syndrome
Brief Title: The Metabolic Effects of Different Weight Loss Diets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNE 595-0107
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Metabolic Syndrome X; Obesity; Insulin Resistance; Hypertension; Diabetes
Keywords: Weight loss; Obesity; Metabolic Syndrome; Diet; Hypertension; Diabetes; Cholesterol
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Insulin Resistance; Hypertension; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Average American Diet (Active Comparator)
  Interventions: Behavioral: Reduced calorie American Diet
- The DASH diet (Active Comparator)
  Interventions: Behavioral: The DASH diet
- The Low Glycemic Index Diet (Active Comparator): The carbohydrate content of a low GI diet can vary, but many advocates of low GL popular diets suggest a macronutrient profile that is 40% carbohydrate, 30% protein, and 30% fat. These low GL diets are lower in carbohydrate content and higher in protein content than the average American diet. Low GL diets typically contain ample amounts of fruits and vegetables, moderate quantities of nuts, legumes, lean meats, fish, and reduced-fat dairy products, and scant amounts of refined grains, potatoes, and sweets
  Interventions: Behavioral: The low glycemic Index Diet

INTERVENTIONS:
Behavioral: The DASH diet — The DASH diet was originally conceived as the optimal diet for individuals with hypertension, based on epidemiologic and clinical trial data suggesting a beneficial effect of plant-based diets on blood pressure It is a diet rich in fruits, vegetables, whole grains, and low-fat dairy products, with moderate amounts of nuts, legumes, fish, and poultry. Consumption of red meat, sweets, and sugary beverages is limited. As a result, the DASH diet contains more potassium, magnesium, calcium, and fiber and less total fat, saturated fat, cholesterol, simple sugars, and sodium than the average American diet
  Arms: The DASH diet
Behavioral: The low glycemic Index Diet — The carbohydrate content of a low GI diet can vary, but many advocates of low GL popular diets suggest a macronutrient profile that is 40% carbohydrate, 30% protein, and 30% fat. These low GL diets are lower in carbohydrate content and higher in protein content than the average American diet. Low GL diets typically contain ample amounts of fruits and vegetables, moderate quantities of nuts, legumes, lean meats, fish, and reduced-fat dairy products, and scant amounts of refined grains, potatoes, and sweets
  Arms: The Low Glycemic Index Diet
Behavioral: Reduced calorie American Diet — The reduced-calorie diets will provide at least the Recommended Daily Allowance (RDA) for protein (0.8 g/kg/day).
  Arms: Average American Diet

SUMMARY:
Current estimates suggest that 65% of American adults are overweight or obese. Excess body weight has been associated with an increased risk of a number of metabolic abnormalities, including high blood sugar, high blood pressure, high triglyceride levels, and low HDL ("good") cholesterol levels. Insulin resistance (when the body becomes less sensitive to the blood sugar-lowering hormone insulin, and more of the hormone is needed to keep blood sugar levels under control) also frequently occurs as a result of excess body weight. These abnormalities can all increase the risk of heart disease and other serious medical problems. Individuals who are overweight often have a number of these abnormalities at the same time, a situation which is often called "the metabolic syndrome." Dietary changes, physical activity, and weight loss can lead to improvements in each of the metabolic abnormalities described above. However, the best type of diet for people with the metabolic syndrome is not known. This study has been designed to test the effects of several promising dietary patterns, with and without weight loss, in overweight adults with the metabolic syndrome. Most individuals who have the metabolic syndrome do not know they have the condition, so we will be screening many healthy overweight volunteers to see if they may be eligible.

DETAILED DESCRIPTION:
BACKGROUND:

Several dietary approaches, including the Dietary Approaches to Stop Hypertension study diet (the DASH diet) and the low glycemic index diet (low GI diet), may be helpful for overweight individuals who have the metabolic syndrome. The DASH diet is rich in fruits, vegetables, whole grains, and low-fat dairy products. It also contains moderate amounts of nuts, beans, fish, and poultry. Consumption of red meat, sweets, and sugary beverages is limited. As a result, the DASH diet contains more potassium, magnesium, calcium, and fiber and less total fat, saturated fat, cholesterol, simple sugars, and sodium than the average American diet. The DASH diet has been shown to lower blood pressure and LDL cholesterol ("bad" cholesterol). It has also been shown to be an effective diet for weight loss. It may also reduce inflammation and insulin resistance, two important features of the metabolic syndrome.

Low GI diets are typically lower in carbohydrate content and higher in protein content than the average American diet. Many popular diet books promote the use of low glycemic index diets. In this study, the low GI diet will contain plenty of fruits and vegetables and moderate amounts of nuts, beans, lean meats, fish, and reduced-fat dairy products. Refined grains, potatoes, and sweets will be avoided. The low GI diet can help improve levels of blood sugar and insulin in the blood after meals. It may also help control hunger after meals. Some researchers believe it may promote more weight loss than other diets, especially in people with the metabolic syndrome. The low GI diet may also reduce cholesterol and triglyceride levels.

Although both the DASH diet and the low GI diet appear to have beneficial effects, it is not clear whether one diet is better than the other for people with the metabolic syndrome. It is also not clear whether these diets would be better for weight loss than a reduced-calorie average American diet. This weight loss study has been designed to test the metabolic effects of the DASH diet and the low GI diet, as compared to the average American diet.

STUDY OVERVIEW:

Up to 18 research volunteers will be studied at Rockefeller University Hospital during a multi-phase study of almost 15 weeks duration. This study includes a 2-week run-in period at home, a 19-day inpatient period during which weight will be kept stable, an 8-week outpatient weight loss period, and a 2-week inpatient period of weight stability at a lower body weight. All food will be provided for about 13 weeks (during the inpatient periods and the 8-week outpatient weight loss period). Volunteers will first undergo testing (described below) at baseline, on an average American diet. They will then be randomized to one of three diets (the DASH diet, the low GI diet, or the average American diet). Weight will initially be kept stable for two weeks on the study diet. At the end of the first inpatient period, volunteers will undergo repeat testing to assess the metabolic effects of the diets, in the absence of weight loss. Volunteers will then be discharged to home for 8 weeks, during which they will receive a 50% reduced-calorie study diet. Volunteers will return to Rockefeller University Hospital twice a week during the outpatient phase for weight-management skills training and follow-up with study staff. It is expected that volunteers will lose between 5 and 9% of their starting weights during this time. At the end of the weight loss phase, volunteers will be readmitted to the research hospital for a final 2-week stay. Body weight will be maintained at the new, lower weight, and volunteers will undergo repeat testing on the study diet. At the conclusion of testing, volunteers will be discharged from the hospital and the study will conclude.

TESTING:

During this study, a number of tests and procedures will be performed at various times. These will include:

* Questionnaires about physical activity, eating habits, attitudes about food, quality-of-life, and hunger
* A 3-day record of food intake at baseline
* Use of a pedometer (step-counter) to assess usual physical activity
* Blood tests (including blood sugar, insulin levels, cholesterol levels, fat hormones, and inflammatory markers)
* 24-hour ambulatory blood pressure monitoring
* Measurement of energy expenditure (the rate at which a body burns calories)
* Noninvasive assessment of body composition before and after weight loss
* Insulin clamp procedures (during which insulin and sugar are infused through a vein to help determine how sensitive a person's body is to insulin)

ELIGIBILITY:
Inclusion Criteria:

* Nonsmoking men and premenopausal women, ages 18-45
* Body mass index ≥ 27 kg/m2
* Body weight < 200 kg
* Evidence of insulin resistance, as suggested by any one of the following:
* Fasting glucose ≥ 100 mg/dL
* Impaired glucose tolerance, with a glucose concentration of ≥ 140 mg/dL 2 hours after a 75-gram oral glucose challenge
* A fasting insulin concentration ≥ 9 mIU/L
* At least two of the following:
* Waist circumference > 35" in women or > 40" in men
* Prehypertension or hypertension, with BP > 120/80 mmHg but < 145/90 mmHg on 2 antihypertensive agents or less
* TG > 150 but < 500 mg/dL
* HDL < 40 mg/dL in men or < 50 mg/dL in women
* Willingness to consume only study food and drink for the duration of the study and to be randomized to one of the three diets
* Willingness to maintain consistent intake of coffee and/or tea during the inpatient periods
* Willingness to avoid the use of all over-the-counter or prescription vitamins, dietary supplements, and herbal products during the study, with the exception of the multivitamin supplement (Flintstones® Plus Iron.)
* Willingness to continue current antihypertensive medications at the same dose and schedule throughout the study, unless a change is advised.
* Willingness to avoid the use of non-steroidal anti-inflammatory drugs including low-dose daily aspirin, for at least ten days prior to the first admission and during each admission.
* Willingness to avoid the use of acetaminophen (Tylenol) and furosemide (Lasix) for at least 48 hours prior to and during the 24-hour urine collection.
* Willingness to avoid the use of sulfonamide antibiotics for at least 1 week prior to and during the 24-hour urine collection.

Exclusion Criteria:

* Current tobacco smoking
* History of a bleeding disorder
* Findings suggestive of cardiovascular disease.
* Blood pressure ≥ 145/90 mmHg after 10 minutes of rest on two or more screening visits, or treatment with three or more antihypertensive agents at any blood pressure.
* Fasting glucose ≥ 165 mg/dL, glycosylated hemoglobin > 8%, or any treatment with oral hypoglycemic agents, insulin sensitizing agents , insulin, incretin mimetics, amylin analogues, or endocannabinoid receptor antagonists.
* History of chronic glucocorticoid use, oral glucocorticoid use for more than 5 days in the previous year, or anticipated treatment with oral or intravenous glucocorticoids during the study period.
* Current treatment with weight loss medications.
* History of bariatric surgery
* Current treatment with any cholesterol-lowering medications.
* Hyperthyroidism or untreated hypothyroidism.
* Pregnancy, desired pregnancy, or lactation within the study period.
* Peri- or postmenopausal status.
* Obstructive sleep apnea.
* Active gallstone disease
* Known history of chronic hepatitis, or liver enzymes more than 2.5 times the upper limit of normal
* Known infection with HIV or confirmed positive test for HIV antibody
* Inflammatory bowel disease, active cancer, or any other medical condition that may cause significant acute weight loss or gain
* Sustained weight loss > 5% of body weight in the previous two months, or sustained weight loss > 10% of body weight in the previous six months
* History of kidney stones
* Renal disease, as evidenced by a serum creatinine above the normal limit on more than one screening visit
* Serum calcium, potassium, or magnesium above the normal limit, confirmed on two screening tests
* Seizure disorder
* History of any inpatient psychiatric admission within the past two years
* History of schizophrenia, psychosis, or bipolar disorder
* History of anorexia nervosa or bulimia nervosa or a history of medical or psychological treatment for an eating disorder
* Severe binge eating disorder
* Active moderate to severe depression.
* History of alcohol or drug abuse within the previous two years
* History, physical, or laboratory findings suggestive of any other medical or psychological condition that would, in the opinion of the principal investigator, make the candidate ineligible for the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity over time | Baseline, Inpatient Days 1-19, Inpatient final 2 weeks

SECONDARY OUTCOMES:
Change in body weight | Baseline, Outpatient 2 weeks, inpatient 1-19 days, outpatient 8 weeks and inpatient 2 weeks
Change in blood sugar levels | baseline and final inpatient 2 weeks
Change in blood pressure | Baseline, Inpatient days 1-19 and inpatient 2 weeks
Change in cholesterol levels | Baseline and outpatient 8 weeks
Change in inflammatory markers | Baseline, Inpatient days 1-19 and outpatient 2 weeks
Diet satisfaction | day 88

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Neff, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States